CLINICAL TRIAL: NCT00350935
Title: Attention and Grouping of Visual Information: What is Disturbed in Patients With Schizophrenia?
Brief Title: Attention and Visual Perception in Schizophrenia: A Functional Magnetic Resonance Imaging (fMRI) Study
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Centre National de la Recherche Scientifique, France (Other); Région Alsace (Unknown); Faculté de Médecine de Strasbourg (Unknown)
Responsible Party: Emmanuel LAVOUE, Directeur Adjoint de la DRCI, University Hospital, Strasbourg, France
Other Study IDs: 3456
Record Dates: First submitted 2006-07-10; First posted 2006-07-11 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2010-06

CONDITIONS: Schizophrenia
Keywords: fMRI; Visual perception; Attention
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Healthy volunteers: Healthy controls
  Interventions: Procedure: fMRI
- Patients: Patients with schizophrenia
  Interventions: Procedure: fMRI

INTERVENTIONS:
Procedure: fMRI — One 30 minute session

SUMMARY:
The main objective of the study is to contribute to a better understanding of the physiopathology of schizophrenia, by studying causal relationships between cognitive deficits and the neurobiological basis for these deficits. Processing visual information involves both automatic grouping processes and control processes. Automatic grouping processes allow the building of a global configuration from local contour information. It is necessary in order to recognize objects. Control processes allow tending to and prioritizing information parts. The paradigm the investigators use allows to dissociate these processes, and is used in order to characterize the impairments observed in patients with schizophrenia. It is adapted to fMRI in order to explore the neurobiological basis of the deficits. The investigators will examine whether functional disconnectivity between activated areas subtend the impairments observed in patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with schizophrenia (DSM-IV criteria)
* Healthy controls matched with patients on age, sex and education level
* Ages 18 to 50
* Signed informed consent
* Right-handed

Exclusion Criteria:

* No severe somatic illness
* No invalidating sensory disease
* No drug abuse, as defined by DSM-IV criteria
* No general anaesthesia in the past 3 months
* No intake of drugs affecting the CNS, except for patients

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Primary care clinic, residents of Strasbourg
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2006-09; Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Giersch, MD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Inserm U666 - Département de Psychiatrie, Hôpitaux Universitaires de Strasbourg, Strasbourg, France